CLINICAL TRIAL: NCT07329803
Title: Pre-cut Versus Intentional Double Guidewire for ERCP Cannulation: Prospective, Randomized Controlled Trial
Acronym: PRIDE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterology, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRIDE
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: ERCP; Choledocholithiasis; Biliary Drainage; Biliary Strictures Caused by Malignant Neoplasms; Biliary Stricture
Keywords: Selective CBD cannulation; Post ERCP Pancreatitis; Precut Sphincterotomy; Double Guidewire Technique
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precut Sphincterotomy Arm (Experimental): Participants undergo biliary cannulation using precut sphincterotomy as the initial rescue cannulation technique during ERCP.
  Interventions: Procedure: Double Guidewire Technique
- Double Guidewire Technique Arm (Active Comparator): Participants undergo biliary cannulation using the double guidewire technique, with placement of a guidewire in the pancreatic duct followed by attempted biliary cannulation during ERCP.
  Interventions: Procedure: Precut Sphincterotomy

INTERVENTIONS:
Procedure: Precut Sphincterotomy — Precut sphincterotomy is an endoscopic rescue cannulation technique in which a needle-knife or similar cutting instrument is used to incise the papillary or periampullary tissue to facilitate access to the bile duct during ERCP.
  Arms: Double Guidewire Technique Arm
Procedure: Double Guidewire Technique — The double guidewire technique is an endoscopic rescue cannulation method in which a guidewire is placed into the pancreatic duct to stabilize the papilla, followed by attempted biliary cannulation alongside the pancreatic duct guidewire during ERCP.
  Arms: Precut Sphincterotomy Arm

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an indispensable therapeutic procedure in the management of a wide spectrum of pancreaticobiliary disorders, including choledocholithiasis, benign and malignant biliary strictures, pancreatic ductal obstructions, and postoperative bile leaks. The procedure has revolutionized the management of these conditions, often obviating the need for surgery.Precut papillotomy and Double Guidewire Technique (DGT) are both salvage techniques used in ERCP when standard biliary cannulation fails.

Precut (Needle-Knife Precut): An endoscopic incision made into the papilla to gain access to the bile duct when conventional methods fail.

Intentional Double Guidewire Technique (DGT): A technique where a guidewire is intentionally placed into the pancreatic duct to act as a "guide" or anchor, straightening the biliary axis and allowing a second guidewire to be inserted into the bile duct.

ELIGIBILITY:
Inclusion Criteria:

- Age > 18 years.

* Valid indication for ERCP (benign or malignant obstruction).
* Native papilla (no prior sphincterotomy).
* Difficult Biliary Cannulation (DBC) defined by ESGE "5-5-2" criteria:
* > 5 minutes of cannulation attempts.
* > 5 contacts with the papilla.
* > 1 inadvertent pancreatic duct cannulation.

Exclusion Criteria:

* Ampullary mass or tumor preventing standard cannulation view.

  * Surgically altered anatomy (e.g., Billroth II, Roux-en-Y).
  * Uncorrectable coagulopathy (INR > 1.5 or Platelets < 50,000).
  * Acute pancreatitis present prior to ERCP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Safe Success | 30 Days
  SUCCESS: Deep cannulation of the Common Bile Duct (CBD) achieved using the randomized technique within 15 minutes.
  * AND ABSENCE OF Post ERCP adverse events.
  Post ERCP adverse events include Post ERCP Pancreatitis, Hemorrhage, cholangitis and perforation.

SECONDARY OUTCOMES:
Incidence of Post-ERCP Pancreatitis | 30 days
  Incidence of post-ERCP pancreatitis, defined as new or worsened abdominal pain with serum amylase or lipase ≥3 times the upper limit of normal at ≥24 hours after ERCP, requiring hospitalization or prolongation of planned admission.
Severity of Post-ERCP Pancreatitis | 30 days
  Severity of post-ERCP pancreatitis classified as mild, moderate, or severe according to the revised Atlanta classification.
Overall ERCP-Related Adverse Events | 30 days
  Incidence of ERCP-related adverse events, including bleeding, perforation, cholangitis, and post-ERCP pancreatitis, graded according to the ASGE lexicon.
Cannulation Time | During the ERCP procedure
  Time required to achieve deep biliary cannulation, measured from insertion of the duodenoscope into the second part of the duodenum to successful deep bile duct cannulation.
Total Procedure Time | During the ERCP procedure
  Total ERCP procedure duration, measured from duodenoscope insertion to scope withdrawal.
Need for Rescue Cannulation Technique | During the ERCP procedure
  Proportion of patients requiring crossover to an alternative rescue cannulation technique after failure of the initially assigned technique.
Hyperamylasemia Without Clinical Pancreatitis | At 24 hours after ERCP
  Incidence of asymptomatic hyperamylasemia, defined as serum amylase or lipase ≥3 times the upper limit of normal without clinical features of pancreatitis.
Hospital Length of Stay | Up to 30 days after ERCP
  Duration of hospital stay measured in days from ERCP to hospital discharge
30-Day All-Cause Readmission | Up to 30 days after ERCP
  Rate of hospital readmission for any cause after ERCP.

CONTACTS AND LOCATIONS:
Overall Officials: DR SHUJAATH ASIF, MD,DM, Principal Investigator — Asian Institute Of Gastroenterology Private Limited

IPD SHARING:
Plan to Share IPD: No